CLINICAL TRIAL: NCT07074379
Title: Endotherapy and/or Extracorporeal Shockwave Lithotripsy Versus Conservative Treatment in Painless Chronic Pancreatitis
Brief Title: Endotherapy and/or Extracorporeal Shockwave Lithotripsy for Painless Chronic Pancreatitis
Acronym: PCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCP
Record Dates: First submitted 2025-06-29; First posted 2025-07-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Painless Chronic Pancreatitis
MeSH Terms: interventions — Metformin; Insulin; Cholangiopancreatography, Endoscopic Retrograde; Lithotripsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotherapy and/or Extracorporeal Shockwave Lithotripsy Group (Experimental): Participants in this arm will undergo a comprehensive treatment approach that includes lifestyle modifications, pharmacological interventions, and procedural therapies such as endoscopic retrograde cholangiopancreatography (ERCP) and/or extracorporeal shockwave lithotripsy (ESWL).
  Interventions: Behavioral: Lifestyle modifications; Drug: Pancreatic enzyme (Pancreatin Enteric-coated Capsules or Oryz-Aspergillus Enzyme and Pancreatin Table), antidiabetic medicine(Acarbose , Metformin, Glimepirde Tablets, Insulin); Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP) and/or Extracorporeal Shockwave Lithotripsy (ESWL)
- Conservative Treatment Group (Active Comparator): This arm includes participants who will receive standard conservative management for painless chronic pancreatitis. The treatment regimen comprises lifestyle modification and medications to manage symptoms of pancreatic exocrine and endocrine insufficiency, such as pancreatic enzyme supplements and medications for diabetes management (e.g., oral hypoglycemics or insulin).
  Interventions: Behavioral: Lifestyle modifications; Drug: Pancreatic enzyme (Pancreatin Enteric-coated Capsules or Oryz-Aspergillus Enzyme and Pancreatin Table), antidiabetic medicine(Acarbose , Metformin, Glimepirde Tablets, Insulin)

INTERVENTIONS:
Behavioral: Lifestyle modifications — Lifestyle modifications primarily include quitting smoking and alcohol consumption, as well as engaging in physical exercise.
Drug: Pancreatic enzyme (Pancreatin Enteric-coated Capsules or Oryz-Aspergillus Enzyme and Pancreatin Table), antidiabetic medicine(Acarbose , Metformin, Glimepirde Tablets, Insulin) — This intervention involves the use of medications to control the pancreatic exocrine and endocrine dysfunction caused by chronic pancreatitis.
  1. Pancreatic enzyme therapy: Patients will use pancreatic enzymes (pancreatin enteric-coated capsules or oryz-aspergillus enzyme and pancreatin tablets) to control the symptoms of exocrine pancreatic insufficiency.
  2. Diabetes treatment: Patients with diabetes will also use antidiabetic medications (such as oral hypoglycemic drugs or insulin, depending on glycemic control needs).
Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP) and/or Extracorporeal Shockwave Lithotripsy (ESWL) — This intervention involves the application of endoscopic retrograde cholangiopancreatography (ERCP) and/or extracorporeal shockwave lithotripsy (ESWL), conducted in accordance with established clinical guidelines. The procedures are tailored to the individual patient's condition, which may include sphincterotomy, balloon dilation of pancreatic duct strictures, stone extraction, and stent placement as indicated. ESWL may be used prior to ERCP to fragment pancreatic duct stones, facilitating their removal.
  Arms: Endotherapy and/or Extracorporeal Shockwave Lithotripsy Group

SUMMARY:
Chronic pancreatitis (CP) is caused by factors such as genetics and the environment, leading to the destruction of pancreatic tissue, infiltration of inflammatory cells, and progressive fibrosis of the pancreas. As the disease progresses, pancreatic tissue is damaged, resulting in impaired endocrine and exocrine functions, manifesting as symptoms like steatorrhea and diabetes. Pain associated with chronic pancreatitis (PACP) is the most common symptom in CP patients. Approximately 75% of patients initially present with abdominal pain, and previous studies have shown that PACP can occur in 85-97% of CP patients. However, there is a type of pancreatitis where patients do not experience abdominal pain and typically seek medical attention due to routine check-ups or symptoms of pancreatic endocrine and exocrine dysfunction; this particular type of pancreatitis is known as painless CP. A meta-analysis showed that painless CP accounts for about 12% of all CP patients.

In patients with CP, continuous pancreatic damage leads to the destruction of pancreatic tissue, subsequently causing insufficiency in both exocrine and endocrine functions. "Painless" does not equate to "harmless"; patients with painless CP often present with severe symptoms of pancreatic exocrine and endocrine dysfunction at the time of diagnosis. These findings underscore the importance of early identification and active management of patients with painless CP.

Whether active endoscopic intervention is needed for painless CP remains a matter of debate. The European Society of Gastrointestinal Endoscopy (ESGE) suggests endoscopic therapy and/or extracorporeal shockwave lithotripsy (ESWL) as the first-line therapy for painful uncomplicated chronic pancreatitis (CP) with an obstructed main pancreatic duct (MPD) in the head/ body of the pancreas; however, due to the unclear potential benefits (preservation of pancreatic function) of endoscopic and/or ESWL treatment for painless CP, it is not recommended for patients without pain, although the evidence is of low quality.

Although there is currently no consensus on whether endoscopic treatment can protect the pancreatic function of patients with painless chronic pancreatitis, preliminary evidence suggests that endoscopic treatment may have a positive impact on pancreatic atrophy and dysfunction in patients with painless CP. In a retrospective study by Ikeura et al., which included 268 patients with CP and painless pancreatic duct stones, it was found that endoscopic treatment and complete clearance of stones in patients with painless pancreatic duct stones helped maintain the volume of the pancreatic parenchyma.

Although preliminary research suggests that endoscopic treatment may protect pancreatic function in patients with painless CP, it could also trigger pain. A study by Ikeura et al. found that painless CP patients who underwent endoscopic treatment but did not have complete clearance of pancreatic duct stones were at a significantly higher risk of developing pain. This indicates that incomplete endoscopic treatment might lead patients from a painless state to one of pain. However, a study by Amodio et al. suggests that the likelihood of painless CP patients experiencing pain in the short term is low, implying that conservative treatment might be more appropriate.

Current research on the clinical characteristics of painless CP and its response to treatment is relatively limited, necessitating further clinical studies to clarify the impact of ERCP and/or ESWL on these patients. We plan to conduct a randomized controlled trial to assess whether these minimally invasive interventions can improve clinical outcomes for patients with painless CP

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 years.
* Diagnosed with painless chronic pancreatitis.
* No prior history of endoscopic retrograde cholangiopancreatography (ERCP) or extracorporeal shockwave lithotripsy (ESWL) treatment.

Exclusion Criteria:

* Presence of complications requiring endoscopic or surgical intervention, such as pancreatic pseudocysts, benign biliary strictures, or pancreatic fistulas.
* Autoimmune pancreatitis.
* Suspected malignancy.
* History of pancreatic surgery or gastrointestinal bypass surgery (e.g., Billroth II procedure).
* End-stage disease.
* Pregnancy or lactation.
* Contraindications to ESWL or ERCP.
* Refusal to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Acute Pancreatitis Incidence | 12 months
  The incidence of acute pancreatitis assessed by Revised Atlanta Classification over a 12-month period following randomization.

SECONDARY OUTCOMES:
Severity of Acute Pancreatitis | 12 months
  The severity of acute pancreatitis episodes that occur within 12 months post randomization. Severity will be graded according to the Atlanta Classification criteria, which categorizes pancreatitis into mild, moderate, and severe based on clinical and imaging findings.
Incidence and Severity of Pancreatic Pain | 12 months
  The incidence and severity of pancreatic pain over a 12-month period. Pain severity will be measured using the Visual Analogue Scale (VAS), where patients rate their pain on a scale from 0 (no pain) to 10 (worst possible pain).
Pancreatic Exocrine Function | 12 months
  This outcome assesses changes in pancreatic exocrine function by measuring fecal elastase-1 levels at baseline and 12 months post randomization.
Glycosylated Hemoglobin Level | 12 months
  This outcome measure evaluates the percentage of hemoglobin that is glycosylated, reflecting the average blood glucose levels over the past 2 to 3 months. It is a key indicator of long-term glycose level in patients.
Fasting Blood Glucose Level | 12 months
  This outcome measure assesses the level of glucose in the blood after an overnight fast. Fasting glucose is a standard test for diagnosing diabetes and monitoring diabetes control. It provides a snapshot of the body's ability to manage glucose without the influence of food.
Fasting C-Peptide Concentration | 12 months
  This outcome measure determines the concentration of C-peptide in the blood during a fasting state. C-peptide is a byproduct of insulin production and provides an index of endogenous insulin secretion. It is useful for assessing insulin production capacity.
C-peptide Area Under the Curve (AUC) Post MMTT | 12 months
  This outcome measures the total exposure to C-peptide over the first 2 hours following a mixed meal tolerance test (MMTT). The AUC is calculated using Riemann sums based on the midpoint of each interval (0, 30, 60, 90, and 120 minutes). This metric is crucial for assessing the overall insulin secretion capacity of the islets.
Glucose Area Under the Curve (AUC) Post MMTT | 12 months
  This outcome assesses the total glucose exposure over the first 2 hours following a Mixed Meal Tolerance Test (MMTT). The AUC is determined using Riemann sums based on the midpoint of each interval (0, 30, 60, 90, and 120 minutes). This metric is essential for evaluating the body's glucose handling ability and the effectiveness of glucose control.
Insulin Area Under the Curve (AUC) Post MMTT | 12 months
  This outcome measures the total insulin exposure over the first 2 hours following a Mixed Meal Tolerance Test (MMTT). The AUC is calculated using Riemann sums based on the midpoint of each interval (0, 30, 60, 90, and 120 minutes). This metric is vital for assessing the overall insulin secretion response to a meal and the effectiveness of insulin production.
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 12 months
  The HOMA-IR is calculated from fasting glucose and fasting insulin levels obtained during the MMTT. It provides an estimate of insulin resistance and is calculated using the formula: HOMA-IR= (fasting glucose × fasting insulin)/405. This index is crucial for understanding the body's insulin sensitivity.
Homeostatic Model Assessment of β-cell Function (HOMA-b) | 12 months
  HOMA-b is determined by the formula HOMA b = (fasting insulin × 360)/(fasting glucose - 63) to assess insulin secretion. It provides an estimate of the β-cell function in response to fasting glucose levels.
Insulinogenic Index Post MMTT | 12 months
  The insulinogenic index is a measure of the early insulin response to a glucose challenge, calculated as (Δinsulin30-0min / Δglucose30-0min). It reflects the capacity of the β-cells to secrete insulin in response to a rise in blood glucose levels.
C-peptide Secretion Index Post MMTT | 12 months
  This index is calculated by replacing insulin with C-peptide in the insulinogenic index formula, i.e., (ΔC-peptide30-0min / Δglucose30-0min). It serves as a measure of the early C-peptide response to a glucose challenge, providing information about the secretory capacity of the islets.
Disposition Index for C-peptide | 12 months
  The disposition index for C-peptide is calculated as (ΔC-peptide30-0min / Δglucose30-0min) × (1 / fasting C-peptide). It represents the ratio of insulin or C-peptide secretion to sensitivity and is an important indicator of the overall β-cell function and insulin sensitivity.
Quality of Life Assessed by SF-36 | 12 months
  This outcome evaluates the quality of life (QoL) of patients with painless chronic pancreatitis at two time points: at baseline (time of hospital admission) and at 12 months post-randomization. The assessment is conducted using the Short Form Health Survey (SF-36), a widely recognized and validated tool that measures health-related quality of life across eight dimensions: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The SF-36 provides a comprehensive overview of how the condition and treatment affect the patients' overall well-being and daily functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided